CLINICAL TRIAL: NCT04177381
Title: Comparative Study Between Subcutaneous Tissue Closure Versus Drain in Obese Women Undergo Elective Cesarean Section Arandomized Controlled Trial
Brief Title: Comparative Study Between Subcutaneous Tissue Closure Versus Drain in Obese Women Undergo Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 171
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Cesarean Section

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- interrupted closure of subcutaneous tissue with drain (Active Comparator): consist of 89 patients that will be allocated for interrupted closure of subcutaneous tissue with drain
  Interventions: Procedure: Cesarean section; Procedure: subcutanous sutures; Device: subcutanous drain
- interrupted closure of subcutaneous tissue without dra (Active Comparator): consist of 88 patients that will be allocated for interrupted closure of subcutaneous tissue without drain
  Interventions: Procedure: Cesarean section; Procedure: subcutanous sutures
- non closure of subcutaneous tissue with drain (Active Comparator): In the drain group,a closed non vacuum drain will be inserted in the tissue and exit from the skin through a separate opening and stitch to the skin
  Interventions: Procedure: Cesarean section; Device: subcutanous drain
- non closure of subcutaneous tissue and no drain (Active Comparator): 87 women without subcutanous sutures and without drain
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean section — 1. Abdominal Incision: Pfannenstiel incision Sharp dissection will be continued through the subcutaneous layer to the fascia.
  2. The fascia will be then incised sharply at the midline
  3. The transversalis fascia and pre peritoneal fat will be dissected carefully
  4. The peritoneum will be then incised.
  5. Low Transverse Cesarean Incision. Bladder flap creation effectively moves the bladder away from the planned hysterotomy site
  6. Delivery of the Fetus and placenta.
  7. Uterine Repair in two layers of continuous 0-or No.1 absorbable suture.
Procedure: subcutanous sutures — suture closure of subcutaneous tissue with interrupted 2-0 polyglactin 910 (Vicryl).the stitch interval is 1cm
  Arms: interrupted closure of subcutaneous tissue with drain; interrupted closure of subcutaneous tissue without dra
Device: subcutanous drain — Inthedraingroup,aclosednonvacuum drain willbeinsertedin thetissueandexitefrom theskinthroughaseparateopeningandstitchto theskin
  Arms: interrupted closure of subcutaneous tissue with drain; non closure of subcutaneous tissue with drain

SUMMARY:
Randomised cinical trial in Kasr Alainy Hospital.352 obese women pregnant with gestational age >38 wk ,theire age range from (25-35) years and BMI between (30 -40) undergoing elective cesarean section were randomised into 4 groups and compare the role of subcutaneous tissue closure in post cesarean section wound complications.

groups are: 4 groups each group was 86 women : A -interrupted closure of subcutaneous tissue with drain ( a closed nonvacuum drain was inserted in the tissue and exite from the skin through a separate opening and stitch to the skin) .

B-interrupted closure of subcutaneous tissue without drain. c- non closure of subcutaneous tissue with drain only. d- non closure of subcutaneous tissue without drain.

All womenu nder going CS with Pfannenstiel incision were considered to be eligible if time allowed informed consent before the surgery

DETAILED DESCRIPTION:
Randomised cinical trial in Kasr Alainy Hospital.352 obese women pregnant with gestational age >38 wk ,their age range from (25-35) years and BMI between (30 -40) undergoing elective cesarean section were randomised into 3 groups (100 patients in each group)and compare the role of subcutaneous tissue closure in post cesarean section wound complications.

4 groups are:: A -interrupted closure of subcutaneous tissue with drain ( a closed nonvacuum drain was inserted in the tissue and exit from the skin through a separate opening and stitch to the skin) .

B-interrupted closure of subcutaneous tissue without drain. c- non closure of subcutaneous tissue with drain only. d- non closure of subcutaneous tissue without drain.

All women under going CS with Pfannenstiel incision were considered to be eligible if time allowed informed consent before the surgery All surgical procedures were performed by obstetric and gynecology residents under the supervision of attending physicians After the sequential closure of the uterus and peritoneum, the fascia was closed with 2-0 polyglactin 910 (Vicryl). The depth of the subcutaneous adipose tissue was measured with a sterile ruler from the fascia to the skin edge at the middle of the superior aspect of the skin incision.Women with a subcutaneous tissue thickness of 4.0 cm or more were then formally enrolled and randomized to one of the two subcutaneous closure techniques. Subcutaneous hemostasis were achieved using electrocautery and skin was approximated with subcuticular suture using 2-0 polyglactin910 (VicrylRapide).company city country In the drain group, a closed nonvacuum drain was inserted in the tissue and exite from the skin through a separate opening and stitch to the skin (Al Allair 2000). company city country The drain was left until the drainage rate was less than 30 ml/day or after 72h .( The skin was closed with a continuous nonabsorbable polypropylene 2/0 (Acufirm; Ernst Kratz, Germany) subcuticular sutures. Operative time was estimated from the start of skin incision until the end of skin suturing. The drain was left until the drainage rate was less than 50 ml/day.

All randomized women received standard postoperative wound care. Surgical dressing was removed on the first postoperative and all participants were discharged 24 h after the CS. The participants were invited to two follow-up in the first and second week post operative with regard to postoperative pain, postoperative fever, hospital stay duration, wound infection, wound seroma, wound disruption, and the need for redressing. The postoperative pain was judged after 24 h using visual analogue scale, in addition any time clinically indicated. Patients and physicians who assessed the incision postoperatively were blinded towards the study group.

ELIGIBILITY:
Inclusion Criteria:

* obese women who BMI(30- 40 kg/m2)
* Gestational age (37-41) week calculated by sure dates and confirmed by first trimester US,
* single fetus.
* Elective lower segment cesarean section

Exclusion Criteria:

* Any medical disorders affect wound healing as:
* Diabetes mellitus.
* On steroids.
* Immunedeficiency.
* Hypoalbuminemia.
* Skin infections or history of wound infections.
* Multifetal pregnancy.
* Obstetric complications eg.placenta previa.
* Anemia.
* Intraoperative complications as intestinal injury or bladder injury

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 352 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
wound infection | 2-8 weeks after the operation
  subjective evaluation of wound redness, seroma and induration

CONTACTS AND LOCATIONS:
Overall Officials: ahmed maged, Study Director — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shalaby MA, Metwally HHM, Maged AM, Bayoumi YA, Salah N. The value of subcutaneous tissue closure and drain in obese women undergo elective caesarean section: a randomized controlled trial. BMC Pregnancy Childbirth. 2025 May 5;25(1):534. doi: 10.1186/s12884-025-07579-z. PMID 40325365